CLINICAL TRIAL: NCT06738381
Title: Individually Tailored Digital Secondary Prevention After Hospitalization for Atherosclerotic Cardiovascular Disease: a Randomized Proof-of-concept Study
Brief Title: Digital Secondary Prevention After Atherosclerotic Cardiovascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 807276
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Atheroscleroses, Coronary; Atheroscleroses, Cerebral; Atherosclerotic Ischemic Disease
MeSH Terms: conditions — Coronary Artery Disease; Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital intervention and motivational counselling (Experimental): A single in-hospital motivational counselling session and access to a digital platform for a 6 months period with patient information, videos and an individualized treatment plan and follow-up plan.
  Interventions: Behavioral: Digital intervention and motivational counselling
- Control group (Active Comparator): Brief advices, tailored discharge information to patients and their general practitioners, and a nurse-led outpatient visit at six months follow-up
  Interventions: Behavioral: Digital intervention and motivational counselling

INTERVENTIONS:
Behavioral: Digital intervention and motivational counselling — A single sesstion of motivational interviewing and access to a digital plattform for a six months period

SUMMARY:
Atherosclerotic cardiovascular disease (ASCVD) remains a leading cause of morbidity and mortality worldwide and in Norway. Approximately 50% of the patients admitted to hospitals with an acute ASCVD event has had a previous event. The high number of patients being readmitted to hospitals with new ASCVD events is to a large degree explained by poor control of established risk factors such as high LDL-cholesterol, high blood pressure (BP), diabetes, obesity, smoking, and lack of physical activity, as well as poor adherence to evidence-based medication. This pragmatic, open-label proof-of-concept study conducted at three secondary care hospitals will randomly assign patients hospitalized with an ASCVD event to either: (i) brief advice, tailored discharge information to general practitioners, and a nurse-led outpatient visit (control), or (ii) the same interventions as (i) plus a single in-hospital motivational counselling session and access to a digital platform for a 6 months period with patient information/videos and an individualized treatment plan and follow-up plan. The primary end point will be between-group differences in the proportion who report having attended follow-up visits in primary (primary care physicians and community-based healthy life centres) and specialist (cardiac rehabilitation programs, hospital outpatient visits) healthcare after 8 weeks and 6 months follow-up. Secondary end points will be change in the SMART2 risk score and cardiovascular risk factors between baseline and 6 and 12 months follow-up. Exploratory end points will be changes in adherence to cardiovascular drugs, self-care behaviour, health literacy, patient activation, and quality of life.

ELIGIBILITY:
Inclusion criteria (all the following):

* Aged >=18 years and signed informed consent and expected cooperation according to ICH/GCP and national/local regulations
* Hospitalised with an planned or unplanned ASCVD event and/or established atherosclerosis
* Access to a smartphone or tablet

Exclusion criteria (any of the following):

-Any condition or situation, that in the investigator's opinion could put the subject at significant risk, confound the study results, interfere significantly with the subject participation in the study, or rendering informed consent unfeasible not limited to: cognitive impairment, seizure disorders, active suicidal intent or plans, substance or alcohol dependence, psychotic disease, major depressive disorders or bipolar disorders, receiving concurrent psychological treatments, and ongoing night shift work.

* Short life expectancy (<12 months) due to end-organ (i.e COPD 4, CKD 4/5) or malignant diseases
* Clinically significant symptoms of anxiety and depression (HADS A and/or HADS-D score ≥8)
* Not being able to understand Norwegian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Attended follow-up visits in primary healthcare | From baseline to weeks 6-8 and 26
  Between-group differences in the proportion attending follow-up visits at primary care physicians and community-based healthy life centres assessed by patient self-report and from medical records
Attended follow-up visits in specialist healthcare | From baseline to weeks 6-8 and 26
  Between-group differences in the proportion attending follow-up visits at cardiac rehabilitation programs and at hospital outpatient visits assessed by patient self-report and from hospital medical records

SECONDARY OUTCOMES:
Change in the SMART2 risk score | From baseline to weeks 26 and 52
  Between-group change in the validated SMART2 risk score
Changes in lipid profile | From baseline to weeks 26 and 52
  Between-group changes in total cholesterol, HDL-cholesterol and LDL-cholesterol in blood
Changes in systolic blood pressure | From baseline to weeks 26 and 52
  Between-group changes in systolic blood pressure
Changes in HbA1c | From baseline to weeks 26 and 52
  Between-group change in HbA1c levels in blood
Changes in smoking status | From baseline to weeks 26 and 52
  Between-group differences in the proportion who report smoking abstinence

CONTACTS AND LOCATIONS:
Locations (1):
- Vestre Viken Trust Drammen hospital, Drammen, Buskerud, Norway